CLINICAL TRIAL: NCT04447885
Title: Weighted Blankets and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Laura Case, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 200628
Record Dates: First submitted 2020-06-18; First posted 2020-06-25 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain; Chronic Pain Syndrome
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental blanket (Experimental): This blanket is the weight being tested which cannot be disclosed without unblinding participants.
  Interventions: Device: weighted blanket
- Control blanket (Active Comparator): This blanket is the control weight which cannot be disclosed without unblinding participants.
  Interventions: Device: weighted blanket

INTERVENTIONS:
Device: weighted blanket — A weighted blanket is a blanket with extra weight sewn in for added pressure to the body.

SUMMARY:
The purpose of the study is to test whether the use of weighted blankets can change the experience of chronic pain and to examine if social, psychological, or health factors influence the perception of the blanket. Multiple blanket weights will be tested.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Fluent in English
3. Diagnosis of chronic pain (self-report; those already indicating this diagnosis on researchmatch.org)
4. Willing to sleep with a weighted blanket and fitness watch for 1 week
5. Able to safely lift up to 15lb
6. Willing and able to use their personal smartphone for fitness tracker app and EMA app to submit ratings using personal data plan

Exclusion Criteria:

1. Pregnancy
2. Major medical conditions such as kidney, liver, cardiovascular (hypertension, preexisting cardiac arrhythmia), autonomic, pulmonary, or neurological problems (e.g., seizure disorder)
3. Current or previous use of a weighted blanket
4. Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Change in pain ratings from before to after brief blanket use | 0 and 15 minutes
  Pain ratings will be compared before and after use of weighted blanket on the following scale: Pain VAS: "No pain" to "Worst pain ever" (higher = worse).
Change in pain ratings from before to after nightly blanket use | at baseline (3 nights) and over 7 nights of use
  Pain ratings will be compared before and after 1 week of nightly use of weighted blanket on the following scale: Pain VAS: "No pain" to "Worst pain ever" (higher = worse).

SECONDARY OUTCOMES:
Change in anxiety ratings from before to after brief blanket use | 0 and 15 minutes; also at baseline (3 nights) and over 7 nights of use
  Anxiety ratings will be compared before and after use of weighted blanket on the following scale: Anxiety VAS: "Extremely anxious" to "Neutral" to "Extremely calm" (higher = better).
Change in ratings of sleep quality from before to after brief blanket use | baseline (3 nights) and over 7 nights of use
  Change in sleep quality from before to after use of weighted blanket will be compared on the following scale: perceived sleep quality VAS: "Extremely poor" to "Neutral" to "Extremely good" (higher = better).
Change in sleep quality measured by fitness watch from before to during week of blanket use | baseline (3 nights) and over 7 nights of use
  Change in sleep quality from before to during use of weighted blanket will be compared by measurement of deep vs light sleep from a fitness watch.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baumgartner JN, Quintana D, Leija L, Schuster NM, Bruno KA, Castellanos JP, Case LK. Widespread Pressure Delivered by a Weighted Blanket Reduces Chronic Pain: A Randomized Controlled Trial. J Pain. 2022 Jan;23(1):156-174. doi: 10.1016/j.jpain.2021.07.009. Epub 2021 Aug 20. PMID 34425251